CLINICAL TRIAL: NCT06047600
Title: Optimization of the Surgical Care Pathway for Kidney Tumors by Digitizing Perioperative Nursing Coordination
Brief Title: Optimization of the Surgical Care Pathway for Kidney Tumors by Digitizing Perioperative Nursing Coordination (UroCCR 126)
Acronym: DiPRU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX2022/77
Record Dates: First submitted 2023-09-06; First posted 2023-09-21 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Digitizing Perioperative Nursing Coordination
Keywords: Kidney tumor; Digital tool; Care pathways; Cost analysis; Health economic evaluation
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: cross-sectional stepped wedge cluster randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group is based on the pre-existing organization, with no digital patient follow-up tools.
- Uroconnect Follow Up Group (Experimental): The UroConnect device has a "patient" interface for presenting self-questionnaires and access to a library of educational content and a "caregiver" interface to rationalize and optimize the nurse's activity of perioperative coordination in his task
  Interventions: Other: Uroconnect Follow Up Group

INTERVENTIONS:
Other: Uroconnect Follow Up Group — Inplementation of UroConnect remote monitoring Medical Device (DM) to optimize patient support and nursing coordination.
  Arms: Uroconnect Follow Up Group

SUMMARY:
The project proposes to evaluate the interest of the UroConnect remote monitoring Medical Device (DM) to optimize patient support and nursing coordination

DETAILED DESCRIPTION:
Kidney cancer represents 2 to 3% of solid cancers in adults. Worldwide, an estimated 431,288 people a year are diagnosed with kidney cancer. Each year, in France, 13,500 patients undergo total or partial nephrectomy. The development of minimally invasive surgical techniques and the structuring of innovative care pathways for the management of renal tumors in Enhanced Rehabilitation After Surgery (RAAC) and even on an outpatient basis have led to a significant reduction in the length of stays. The physiognomy of the course of care for patients operated on for a renal tumor is completely modified and generates for the patient a feeling of deterioration in the quality of care and disruption of medical follow-up.

The objective is to deploy a model for coordinating the perioperative care pathway of patients who have undergone nephrectomy for renal tumor in several French centers in order to assess the impact for patients, caregivers and the health system.

This coordination would lead to the formalization of a nurse coordinator job profile adapted to the specificities of oncological surgery and the tools necessary for its implementation. The UroConnect device has a "patient" interface for presenting self-questionnaires and access to a library of educational content and a "caregiver" interface to rationalize and optimize the nurse's activity of perioperative coordination in his task.

ELIGIBILITY:
Inclusion Criteria:

* Planned surgical management by total or partial nephrectomy for kidney tumor,
* Affiliation or beneficiary of the French social security
* Expressed consent for integration of the UroCCR cohort,
* Expressed consent to participate in the DiPRU study.

Exclusion Criteria:

* Difficulties understanding and expressing oneself in French
* Participant under guardianship or curatorship
* Pregnancy at the time of surgery
* No internet access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1307 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-10-23 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of unscheduled and uncoordinated care utilizations | 30 post-operative days
  In the 30 post-operative days, number of unscheduled and uncoordinated care utilizations (emergency visits, re-hospitalizations in urology, general medicine or urology consultations) corresponding to the difference between the use of care identified in the National health data system (SNDS) and scheduled and coordinated care, identified in the patient file of the initial hospitalization for scheduled care and by the coordinating nurse for coordinated care.

SECONDARY OUTCOMES:
Patient anxiety evaluation | Day-1
  Patient anxiety measured by the State-Trait Anxiety Inventory STAI, The STAI questionnaire assesses anxiety as a personality trait and an emotional state and comprised 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety.
Hospitalised patient satisfaction and experience evaluation | Day-30 post-op
  Patient satisfaction and experience measured by the e-Satis questionnaire .The e-satis questionnaire was created and validated in French by the Haute Autorité de Santé (HAS). It is used as a continuous measure of inpatient satisfaction and experience. It is therefore routinely collected by the HAS.
  the e-Satis questionnaires are divided into "dimensions" of the patient pathway (from admission to discharge). Patients respond on a scale ranging from "poor" to "excellent" or from "never" to "always". For each dimension, an overall patient experience and satisfaction score is calculated (A score calculation guide is available on the HAS website).
Nature and reasons for seeking care | Day 30
  Nature and reasons for seeking care declared by the patient and confirmed by the doctor who treated him/her
Average length of stay | Day 30
  Number of re-hospitalizations for complications at D30, use of medical care (medical consultations and hospitalizations) in the 30 days following surgery (SNDS).
UroConnect usage | Month 24
  Number of alerts generated by UroConnect.
Nursing coordination activity linked to UroConnect | Month 24
  Evaluation of nurse activity due to patient requests on UroConnect
Qualitative analysis of the obstacles and levers to appropriation of UroConnect | Month 24
  In each center, professionals and patients will be asked to take part in an individual interviews. This interview will focus on understanding the determining factors in the appropriation of the system and its impact from the point of view of professionals and patients, by identifying 1/ the factors that hinder and encourage appropriation of the system, 2/ the nature of the changes brought about in professional practice and in the patient's care pathway, the patient's feelings in terms of effects on his or her quality of life, disease management and relationship with carers, 3/ the individual, contextual, sociocultural and technical factors in the effectiveness of the intervention.Interview guides will be drawn up in advance, in line with the objectives and hypotheses of the research, and based on the findings of existing literature, such as theoretical models of behavioral and organizational change.
Differential real cost for the Hospital | Month 24
  Difference in actual costs (€), from the hospital's point of view, between phases with and without the digital tool .
Differential cost-consequence ratio | Day 30
  Difference in inpatient and outpatient costs (€) between the 2 strategies

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU d'Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - Centre Catalan d'Urologie, Cabestany
  - CHU de Caen, Caen
  - Hôpital Henri Mondor, Créteil
  - APHM, Marseille
  - CH de Mont de Marsan, Mont-de-Marsan
  - CHU de Nantes, Nantes
  - CHU de Nîmes, Nîmes
  - CHU de Strasbourg, Strasbourg
  - CHu de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided